CLINICAL TRIAL: NCT00408031
Title: N-methyl-D-aspartate Receptor (NMDAR)-Based Pharmacotherapy With D-cycloserine for Treatment-resistant Major Depressive Disorder
Brief Title: D-cycloserine for Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herzog Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Heresco-Levi Uriel, Princepal Investigator, Herzog Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Heresco 4 CTIL; Herzog - protocol 5372; NCT00781014 (obsolete NCT alias)
Record Dates: First submitted 2006-12-03; First posted 2006-12-05 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; NMDA receptor; Treatment-Resistant; D-cycloserine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- 1 (Experimental): Randomization to 2 treatment groups. One group receives adjuvant treatment with D-cycloserine, up to 1 g/day. The second group receives adjuvant treatment with placebo, up to 1 g/day.
  Interventions: Drug: D-cycloserine

INTERVENTIONS:
Drug: D-cycloserine — D-cycloserine (DCS , Seromycin) is a broad spectrum antibiotic, in use for over thirty years against tuberculosis, that acts as a partial agonist at the NMDAR-associated GLY site.

SUMMARY:
For many depression patients treatment changes are required, including switching to another antidepressant and addition of a second antidepressant or a non-antidepressant agent ("augmentation"). The need to modify treatment is usually necessary because of partial or no response to first-line monotherapy or the failure to achieve remission although treatment response (improvement) has been obtained. These caveats of presently available antidepressant drugs highlight the need for innovative pharmacological treatment strategies. Recent data suggest that N-methyl-D-aspartate receptor (NMDAR) antagonists and partial agonists at the NMDAR-associated glycine binding site may represent a novel type of antidepressant medications. These types of compounds protect vulnerable neurons against a variety of insults, including stress-induced damage, and may serve to enhance and maintain normal synaptic connectivity. In animal models, these compounds mimic the effects of clinically effective antidepressants. Furthermore, down-regulation of the glycine site of the NMDAR was found to be a common feature of currently used antidepressant medications. D-cycloserine (DCS , Seromycin) is a broad spectrum antibiotic, in use for over thirty years against tuberculosis, that acts as a partial agonist at the NMDAR-associated glycine site. Beneficial antidepressant effects have been reported with 500-1000 mg/day DCS regimens in depressed tuberculosis patients and recent preliminary findings suggest that DCS may also be beneficial in the treatment of major depressive disorder. The antidepressant effects of DCS seem to reflect consequences of its capacity to reduce NMDAR receptor function. In the present project, it is proposed to assess, using a random assignment, parallel-group, double blind, placebo controlled design, the effects of a NMDAR -antagonist DCS dose regimen, 250 --> 1000 mg/day for 6 wks, as adjuvant pharmacotherapy for treatment-resistant major depressive disorder patients. The study methodology includes the assessment of DCS effects upon symptoms profile, neurocognitive tests performance, amino acids serum levels, and brain electrophysiology parameters associated with the prepulse inhibition-startle response paradigm. It is hypothesized that significant beneficial DCS treatment effects will be registered.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of major depression .
* HAMD scale score of ≥20 despite at least two adequate antidepressant treatment trials during the current episode.

Exclusion Criteria:

* Underwent ECT treatment during the 3 months preceding the study.
* Change in psychotropic medications doses during the 3 weeks preceding the study.
* Concurrent unstable medical or neurological illness.
* Patients are judged to be potentially violent towards themselves or others, or have a history of drug/alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in 24 item Hamilton Depression Rating Scale (HAMD) scores. Safety measures: UKU scale, vital signs assessments, laboratory parameters (SMA-20, CBC, UA) | 6 weeks
Change in Hamilton Rating Scale for Anxiety (HAMA) scores. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Heresco-Levy, M.D., Principal Investigator — Ezrath Nashim - Herzog Memorial Hospital
Locations (2):
- Israel (2):
  - Ezrath Nashim - Herzog Memorial Hospital & Community Clinics, Jerusalem
  - Ezrath Nashim - Herzog Memorial Hospital, Jerusalem

REFERENCES:
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411